CLINICAL TRIAL: NCT06309316
Title: The Impact of Person Centred Care (PCC) on Mental Outcome and Work Ability in Graves' Disease - the GRAves CarE (GRACE) PCC Project
Brief Title: The Impact of Person Centred Care (PCC) in Grave's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Grace-PCC
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Graves Disease
Keywords: Person Centred Care; Mental fatigue; cost-effectiveness; self-efficacy; eHealth
MeSH Terms: conditions — Graves Disease; Mental Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Person-centred care (PCC) (Experimental): Intervention PCC:
  In addition to usual care, patients will receive PCC through physical visits, telephone and through a web-based platform for 15-months. The primary outcome is after 3 month (we expect the need of support is largest in the beginning) but the the intervention will continue for the period of care 12-18 months, increasing transferability to regular care.
  Usual care:
  Patients with GD have regular meetings with the endocrinologist during the treatment with anti-thyroid drugs and leave blod sampels. Many patients are on sick leave in the beginning of treatment. If questions occur between meetings, patients contact a service centre and get feed-back from the nurse or physician on duty at Sahlgrenska University Hospital in Gothenburg.
  Interventions: Behavioral: Person-centred care (PCC)
- Usual care (No Intervention): Usual care:
  Patients with GD have regular meetings with the endocrinologist during the treatment with anti-thyroid drugs and leave blod sampels. Many patients are on sick leave in the beginning of treatment. If questions occur between meetings, patients contact a service centre and get feed-back from the nurse or physician on duty at Sahlgrenska University Hospital in Gothenburg.

INTERVENTIONS:
Behavioral: Person-centred care (PCC) — In addition to usual care, patients will receive PCC through physical visits, telephone and through a web-based platform for 15-months. Primary outcome is after 3 month (we expect the need of support is largest in the beginning) but the intervention will continue for the period of care 12-18 months, increasing transferability to regular care.
  Arms: Person-centred care (PCC)

SUMMARY:
Mental fatigue (MF) is prevalent after Graves' disease (GD), which is the most common form of hyperthyroidism. We have reported that 38% of patients, compared to 11% of control subjects, suffer from MF more than 1 year after successfully reversing of their hyperthyroidism and that MF is an entity of its own, separated from MF combined with anxiety or depression. The brain pathophysiology is unknown and there is no medical treatment, which requires patients to simply adapt to the situation. In the new national guideline for hyperthyroidism (Jan 2023), rehabilitation is recommended, but currently rarely offered to these patients. The problem is significant for patients, as illustrated by frequent media appeals. In this project, we hypothesise that person-centred care (PCC), which promotes positive coping strategies and increases self-efficacy by engaging patients as partners in their own care, improves MF, reduces sick leave, and lowers the recurrence rate of GD. In two work packages (WP), we will:

WP1 Evaluate the effect of PCC eHealth intervention (telephone and digital platform) as an add-on to usual care vs usual care alone in a randomized controlled trial (RCT) of 220 patients on self-efficacy, days of sick-leave (composite score as primary outcome), MF, recurrence rate of disease, coping strategies, perceived stress, quality of life (QoL) and personality.

WP2 Investigate the cost-effectiveness of the intervention

Patients with GD have impaired long-term QoL. PCC could improve long-term outcomes of this autoimmune disease and may apply to other patient groups. This is in line with the societal aim to reduce mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* First time Graves' diseases with elevated FT4 and/or FT3 and positive TSH receptor antibody (TRAb)

Exclusion Criteria:

* Patients that cannot attend to the protocol
* Patients with moderate-severe/ severe Graves' eye disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2029-02-25 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Composite score of changes | Change from baseline examined at 3 months follow-up.
  A patient is classified as improved, deteriorated or unchanged:
  A patient is classified as improved if:
  at 3 months increased general self-efficacy by ≥ 5 units and reduced sick leave percentage (or unchanged if no sick-leave at baseline) at 3 months follow-up
  A patient is classified as deteriorated if:
  at 3 months reduced general self-efficacy by ≥ 5 units or increased sick-leave percentage (or unchanged if on full-time sick leave at inclusion) Those who have neither improved or deteriorated are classified as unchanged

SECONDARY OUTCOMES:
General Self-Efficacy Scale (GSE) | Change from baseline examined at 6 weeks follow-up.
  Evaluated by the validated questionnaire General Self-Efficacy. Scores are compared between the intervention and the control group. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General Self-Efficacy Scale (GSE) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire General Self-Efficacy. Scores are compared between the intervention and the control group. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General Self-Efficacy Scale (GSE) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire General Self-Efficacy. Scores are compared between the intervention and the control group. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General Self-Efficacy Scale (GSE) | Change from baseline examined at 15 months follow-up.
  Evaluated by the validated questionnaire General Self-Efficacy. Scores are compared between the intervention and the control group. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Days of sick-leave | Change from baseline examined at 6 weeks follow-up.
  Evaluated sick leave days between the intervention and the control group.
Days of sick-leave | Change from baseline examined at 3 months follow-up.
  Evaluated sick leave days between the intervention and the control group.
Days of sick-leave | Change from baseline examined at 6 months follow-up.
  Evaluated sick leave days between the intervention and the control group.
Days of sick-leave | Change from baseline examined at 15 months follow-up.
  Evaluated sick leave days between the intervention and the control group.
Mental fatigue score | Change from baseline examined at 6 weeks follow-up.
  Scores at the Mental Fatigue Scale are compared between the intervention and the control group. Scores is between 0-42 and higher scores mean more brain fatigue.
Mental fatigue score | Change from baseline examined at 3 months follow-up.
  Scores at the Mental Fatigue Scale are compared between the intervention and the control group. Scores is between 0-42 and higher scores mean more brain fatigue.
Mental fatigue score | Change from baseline examined at 6 months follow-up.
  Scores at the Mental Fatigue Scale are compared between the intervention and the control group. Scores is between 0-42 and higher scores mean more brain fatigue.
Mental fatigue score | Change from baseline examined at 15 months follow-up.
  Scores at the Mental Fatigue Scale are compared between the intervention and the control group. Scores is between 0-42 and higher scores mean more brain fatigue.
Coping Orientations to Problems Experienced (Brief cope) | Change from baseline examined at 6 weeks follow-up.
  Evaluated by the validated questionnaire Brief cope. The Brief COPE is a shorter version of the COPE Inventory composed of 28-items rated on a 4-point ordinal scale that measure 14 subscales of coping style (2-items each). The overall mean is calculated with more than three being worse outcome. Coping strategies are compared between the intervention and the control group.
Coping Orientations to Problems Experienced (Brief cope) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire Brief cope. The Brief COPE is a shorter version of the COPE Inventory composed of 28-items rated on a 4-point ordinal scale that measure 14 subscales of coping style (2-items each). The overall mean is calculated with more than three being worse outcome. Coping strategies are compared between the intervention and the control group.
Coping Orientations to Problems Experienced (Brief cope) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire Brief cope. The Brief COPE is a shorter version of the COPE Inventory composed of 28-items rated on a 4-point ordinal scale that measure 14 subscales of coping style (2-items each). The overall mean is calculated with more than three being worse outcome. Coping strategies are compared between the intervention and the control group.
Coping Orientations to Problems Experienced (Brief cope) | Change from baseline examined at 15 months follow-up.
  Evaluated by the validated questionnaire Brief cope. The Brief COPE is a shorter version of the COPE Inventory composed of 28-items rated on a 4-point ordinal scale that measure 14 subscales of coping style (2-items each). The overall mean is calculated with more than three being worse outcome. Coping strategies are compared between the intervention and the control group.
Perceived Stress Scale (PSS-14) | Change from baseline examined at 6 weeks follow-up.
  Evaluated by the validated questionnaire Perceived Stress Scale (PSS-14). Scores are compared between the intervention and the control group. The total score ranges between 0 and 56, with a higher score indicate more symptoms of stress.
Perceived Stress Scale (PSS-14) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire Perceived Stress Scale (PSS-14). Scores are compared between the intervention and the control group. The total score ranges between 0 and 56, with a higher score indicate more symptoms of stress.
Perceived Stress Scale (PSS-14) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire Perceived Stress Scale (PSS-14). Scores are compared between the intervention and the control group. The total score ranges between 0 and 56, with a higher score indicate more symptoms of stress.
Perceived Stress Scale (PSS-14) | Change from baseline examined at 15 months follow-up.
  Evaluated by the validated questionnaire Perceived Stress Scale (PSS-14). Scores are compared between the intervention and the control group. The total score ranges between 0 and 56, with a higher score indicate more symptoms of stress.
Personality Assessment Guardian NEO-FFI-3 | Change from baseline examined at 6 weeks follow-up.
  The NEO Five Factor Inventory-3 (NEO-FFI-3) is a measure of the five domains of personality: neuroticism, extraversion, openness to experience, agreeableness, and conscientiousness.
Personality Assessment Guardian NEO-FFI-3 | Change from baseline examined at 3 months follow-up.
  The NEO Five Factor Inventory-3 (NEO-FFI-3) is a measure of the five domains of personality: neuroticism, extraversion, openness to experience, agreeableness, and conscientiousness.
Personality Assessment Guardian NEO-FFI-3 | Change from baseline examined at 6 months follow-up.
  The NEO Five Factor Inventory-3 (NEO-FFI-3) is a measure of the five domains of personality: neuroticism, extraversion, openness to experience, agreeableness, and conscientiousness.
Personality Assessment Guardian NEO-FFI-3 | Change from baseline examined at 15 months follow-up.
  The NEO Five Factor Inventory-3 (NEO-FFI-3) is a measure of the five domains of personality: neuroticism, extraversion, openness to experience, agreeableness, and conscientiousness.
Comprehensive psychopathological rating questionnaire (CPRS) | Change from baseline examined at 6 weeks follow-up.
  Evaluated by the validated questionnaire the Comprehensive Psychopathological Rating Scale (CPRS). Scores are compared between the intervention and the control group. Higher scores at the Comprehensive Psychopathological Rating Scale mean more symptoms of anxiety and depression. The Scores for anxiety is between 0-27 and for depression is between 0-27.
Comprehensive psychopathological rating questionnaire (CPRS) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire the Comprehensive Psychopathological Rating Scale (CPRS). Scores are compared between the intervention and the control group. Higher scores at the Comprehensive Psychopathological Rating Scale mean more symptoms of anxiety and depression. The Scores for anxiety is between 0-27 and for depression is between 0-27.
Comprehensive psychopathological rating questionnaire (CPRS) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire the Comprehensive Psychopathological Rating Scale (CPRS). Scores are compared between the intervention and the control group. Higher scores at the Comprehensive Psychopathological Rating Scale mean more symptoms of anxiety and depression. The Scores for anxiety is between 0-27 and for depression is between 0-27.
Comprehensive psychopathological rating questionnaire (CPRS) | Change from baseline examined at 15 months follow-up.
  Evaluated by the validated questionnaire the Comprehensive Psychopathological Rating Scale (CPRS). Scores are compared between the intervention and the control group. Higher scores at the Comprehensive Psychopathological Rating Scale mean more symptoms of anxiety and depression. The Scores for anxiety is between 0-27 and for depression is between 0-27.
Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39) | Change from baseline examined at 6 weeks follow-up.
  Evaluated by the validated questionnaire Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39). Scores are compared between the intervention and the control group. ThyPRO scales is scored as a summary score and linearly transformed to range 0- 100. Higher scores at the Thyroid-specific Patient-Reported Outcome short-form means worse quality of life.
Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39). Scores are compared between the intervention and the control group. ThyPRO scales is scored as a summary score and linearly transformed to range 0- 100. Higher scores at the Thyroid-specific Patient-Reported Outcome short-form means worse quality of life.
Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39). Scores are compared between the intervention and the control group. ThyPRO scales is scored as a summary score and linearly transformed to range 0- 100. Higher scores at the Thyroid-specific Patient-Reported Outcome short-form means worse quality of life.
Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39) | Change from baseline examined at 15 months follow-up.
  Evaluated by the validated questionnaire Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39). Scores are compared between the intervention and the control group. ThyPRO scales is scored as a summary score and linearly transformed to range 0- 100. Higher scores at the Thyroid-specific Patient-Reported Outcome short-form means worse quality of life.
Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). | Change from baseline examined at 6 weeks follow-up
  Evaluated by the validated questionnaire the Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). Scores are compared between the intervention and the control group. The range of each score is from 0 to 100, higher scores indicating better health.
Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). | Change from baseline examined at 3 months follow-up
  Evaluated by the validated questionnaire the Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). Scores are compared between the intervention and the control group. The range of each score is from 0 to 100, higher scores indicating better health.
Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). | Change from baseline examined at 6 months follow-up
  Evaluated by the validated questionnaire the Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). Scores are compared between the intervention and the control group. The range of each score is from 0 to 100, higher scores indicating better health.
Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). | Change from baseline examined at 15 months follow-up
  Evaluated by the validated questionnaire the Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). Scores are compared between the intervention and the control group. The range of each score is from 0 to 100, higher scores indicating better health.
EuroQol- health questionnaire (EQ-5D) | Change from baseline examined at 6 weeks follow-up
  Evaluated by the validated questionnaire EuroQol- health (EQ-5D). Scores are compared between the intervention and the control group. Each question may have 1 of 3-level answers, and a visual analog scale (VAS) on which patients can mark their current health state. The EQ-5D-3L index is calculated by subtracting the values of the descriptive EQ-5D system from the numerical value 1. This corresponds to the best possible health status, while an index value of <0 represents the worst possible health status.
EuroQol- health questionnaire (EQ-5D) | Change from baseline examined at 3 months follow-up
  Evaluated by the validated questionnaire EuroQol- health (EQ-5D). Scores are compared between the intervention and the control group. Each question may have 1 of 3-level answers, and a visual analog scale (VAS) on which patients can mark their current health state. The EQ-5D-3L index is calculated by subtracting the values of the descriptive EQ-5D system from the numerical value 1. This corresponds to the best possible health status, while an index value of <0 represents the worst possible health status.
EuroQol- health questionnaire (EQ-5D) | Change from baseline examined at 6 months follow-up
  Evaluated by the validated questionnaire EuroQol- health (EQ-5D). Scores are compared between the intervention and the control group. Each question may have 1 of 3-level answers, and a visual analog scale (VAS) on which patients can mark their current health state. The EQ-5D-3L index is calculated by subtracting the values of the descriptive EQ-5D system from the numerical value 1. This corresponds to the best possible health status, while an index value of <0 represents the worst possible health status.
EuroQol- health questionnaire (EQ-5D) | Change from baseline examined at 15 months follow-up
  Evaluated by the validated questionnaire EuroQol- health (EQ-5D). Scores are compared between the intervention and the control group. Each question may have 1 of 3-level answers, and a visual analog scale (VAS) on which patients can mark their current health state. The EQ-5D-3L index is calculated by subtracting the values of the descriptive EQ-5D system from the numerical value 1. This corresponds to the best possible health status, while an index value of <0 represents the worst possible health status.
Frenchay Activities Index (FAI) | Change from baseline examined at 6 weeks follow-up
  Evaluated by the validated Frenchay Activities Index (FAI). Compare function and work ability between the intervention and the control group. Questionnaire consisting of 15 items on frequency of social everyday activities and the score is based on the frequency with which an activity has been performed during the previous 3 or 6 months. The total score ranges from 0 (inactive) to 45 (very active).
Frenchay Activities Index (FAI) | Change from baseline examined at 3 months follow-up
  Evaluated by the validated Frenchay Activities Index (FAI). Compare function and work ability between the intervention and the control group. Questionnaire consisting of 15 items on frequency of social everyday activities and the score is based on the frequency with which an activity has been performed during the previous 3 or 6 months. The total score ranges from 0 (inactive) to 45 (very active).
Frenchay Activities Index (FAI) | Change from baseline examined at 6 months follow-up
  Evaluated by the validated Frenchay Activities Index (FAI). Compare function and work ability between the intervention and the control group. Questionnaire consisting of 15 items on frequency of social everyday activities and the score is based on the frequency with which an activity has been performed during the previous 3 or 6 months. The total score ranges from 0 (inactive) to 45 (very active).
Frenchay Activities Index (FAI) | Change from baseline examined at 15 months follow-up
  Evaluated by the validated Frenchay Activities Index (FAI). Compare function and work ability between the intervention and the control group. Questionnaire consisting of 15 items on frequency of social everyday activities and the score is based on the frequency with which an activity has been performed during the previous 3 or 6 months. The total score ranges from 0 (inactive) to 45 (very active).
Work Productivity and Activity Impairment questionnaire (WPAI). Productivity and Activity Impairment questionnaire (WPAI) | Change from baseline examined at 6 weeks follow-up
  Evaluated by the validated Work Productivity and Activity Impairment questionnaire (WPAI). Compare Work Productivity and Activity between the intervention and the control group.
  Four main outcomes can be generated from the WPAI-GH and expressed in percentages by multiplying the following scores by 100: 1) percent work time missed due to health = Q2/(Q2 + Q4) for those who were currently employed; 2) percent impairment while working due to health = Q5/10 for those who were currently employed and actually worked in the past seven days; 3) percent overall work impairment due to health Q2/(Q2 + Q4) + ((1 - Q2/(Q2 + Q4)) × (Q5/10)) for those who were currently employed; 4) percent activity impairment due to health Q6/10 for all respondents.
Work Productivity and Activity Impairment questionnaire (WPAI). Productivity and Activity Impairment questionnaire (WPAI) | Change from baseline examined at 3 months follow-up
  Evaluated by the validated Work Productivity and Activity Impairment questionnaire (WPAI). Compare Work Productivity and Activity between the intervention and the control group.
  Four main outcomes can be generated from the WPAI-GH and expressed in percentages by multiplying the following scores by 100: 1) percent work time missed due to health = Q2/(Q2 + Q4) for those who were currently employed; 2) percent impairment while working due to health = Q5/10 for those who were currently employed and actually worked in the past seven days; 3) percent overall work impairment due to health Q2/(Q2 + Q4) + ((1 - Q2/(Q2 + Q4)) × (Q5/10)) for those who were currently employed; 4) percent activity impairment due to health Q6/10 for all respondents.
Work Productivity and Activity Impairment questionnaire (WPAI). Productivity and Activity Impairment questionnaire (WPAI) | Change from baseline examined at 6 months follow-up
  Evaluated by the validated Work Productivity and Activity Impairment questionnaire (WPAI). Compare Work Productivity and Activity between the intervention and the control group.
  Four main outcomes can be generated from the WPAI-GH and expressed in percentages by multiplying the following scores by 100: 1) percent work time missed due to health = Q2/(Q2 + Q4) for those who were currently employed; 2) percent impairment while working due to health = Q5/10 for those who were currently employed and actually worked in the past seven days; 3) percent overall work impairment due to health Q2/(Q2 + Q4) + ((1 - Q2/(Q2 + Q4)) × (Q5/10)) for those who were currently employed; 4) percent activity impairment due to health Q6/10 for all respondents.
Work Productivity and Activity Impairment questionnaire (WPAI). Productivity and Activity Impairment questionnaire (WPAI) | Change from baseline examined at 15 months follow-up
  Evaluated by the validated Work Productivity and Activity Impairment questionnaire (WPAI). Compare Work Productivity and Activity between the intervention and the control group.
  Four main outcomes can be generated from the WPAI-GH and expressed in percentages by multiplying the following scores by 100: 1) percent work time missed due to health = Q2/(Q2 + Q4) for those who were currently employed; 2) percent impairment while working due to health = Q5/10 for those who were currently employed and actually worked in the past seven days; 3) percent overall work impairment due to health Q2/(Q2 + Q4) + ((1 - Q2/(Q2 + Q4)) × (Q5/10)) for those who were currently employed; 4) percent activity impairment due to health Q6/10 for all respondents.
Levels of thyroid autoantibodies | Change from baseline examined at 6 weeks follow-up
  Levels of thyroid autoantibodies, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid autoantibodies | Change from baseline examined at 3 months follow-up
  Levels of thyroid autoantibodies, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid autoantibodies | Change from baseline examined at 6 months follow-up
  Levels of thyroid autoantibodies, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid autoantibodies | Change from baseline examined at 15 months follow-up
  Levels of thyroid autoantibodies, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid hormones | Change from baseline examined at 6 weeks follow-up
  Levels of thyroid hormones, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid hormones | Change from baseline examined at 3 months follow-up
  Levels of thyroid hormones, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid hormones | Change from baseline examined at 6 months follow-up
  Levels of thyroid hormones, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid hormones | Change from baseline examined at 15 months follow-up
  Levels of thyroid hormones, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Clinical Activity Score (CAS) | Change from baseline examined at 6 weeks follow-up
  Comparison of Clinical Activity Score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-10 and higher scores mean more eye symptoms.
Clinical Activity Score (CAS) | Change from baseline examined at 3 months follow-up
  Comparison of Clinical Activity Score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-10 and higher scores mean more eye symptoms.
Clinical Activity Score (CAS) | Change from baseline examined at 6 months follow-up
  Comparison of Clinical Activity Score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-10 and higher scores mean more eye symptoms.
Clinical Activity Score (CAS) | Change from baseline examined at 15 months follow-up
  Comparison of Clinical Activity Score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-10 and higher scores mean more eye symptoms.
Severity score | Change from baseline examined at 6 weeks follow-up
  Comparison of Severity score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-29 and higher scores mean more eye symptoms.
Severity score | Change from baseline examined at 3 months follow-up
  Comparison of Severity score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-29 and higher scores mean more eye symptoms.
Severity score | Change from baseline examined at 6 months follow-up
  Comparison of Severity score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-29 and higher scores mean more eye symptoms.
Severity score | Change from baseline examined at 15 months follow-up
  Comparison of Severity score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-29 and higher scores mean more eye symptoms.
Saltin-Grimby Physical Activity Scale (SGPAS) | Change from baseline examined at 6 weeks follow-up
  Physical activity level, 1-4 (4 highest activity level).
Saltin-Grimby Physical Activity Scale (SGPAS) | Change from baseline examined at 3 months follow-up
  Physical activity level, 1-4 (4 highest activity level).
Saltin-Grimby Physical Activity Scale (SGPAS) | Change from baseline examined at 6 months follow-up
  Physical activity level, 1-4 (4 highest activity level).
Saltin-Grimby Physical Activity Scale (SGPAS) | Change from baseline examined at 15 months follow-up
  Physical activity level, 1-4 (4 highest activity level).
Composite score of changes | Change from 6weeks examined at 3 months follow-up.
  A patient is classified as improved, deteriorated or unchanged:
  A patient is classified as improved if:
  at 3 months increased general self-efficacy by ≥ 5 units and reduced sick leave percentage (or unchanged if no sick-leave at baseline) at 3 months follow-up
  A patient is classified as deteriorated if:
  at 3 months reduced general self-efficacy by ≥ 5 units or increased sick-leave percentage (or unchanged if on full-time sick leave at inclusion) Those who have neither improved or deteriorated are classified as unchanged

CONTACTS AND LOCATIONS:
Overall Officials: Helena Filipsson Nyström, Principal Investigator — Sahlgrenska Universitet sjukhus
Locations (1):
- Agneta Lindo, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided